CLINICAL TRIAL: NCT06761079
Title: Comparison of Thoracolumbar Interfascial Plane Block (TLIP-block) and Local Anesthetic Infiltration in Minimally Invasive Spine Surgery: A Randomized Controlled Trial
Brief Title: Comparison of Thoracolumbar Interfascial Plane Block (TLIP-block) and Local Anesthetic (LA) Infiltration in Minimally Invasive Spine Surgery: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Principal Investigator, Sophitnapa Tanasittiboon, Principal Investigator, Queen Savang Vadhana Memorial Hospital, Thailand
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 047/2566
Record Dates: First submitted 2024-12-25; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Percutaneous Pedicular Screw (PPS) Fixation; Minimally Invasive Transforaminal Lumbar Interbody Fusion (MIS TLIF) Surgeries
Keywords: TLIP block; spine surgery; Thoracolumbar interfascial plane block
MeSH Terms: conditions — Popliteal Pterygium Syndrome

STUDY DESIGN:
Intervention Model Description: Patients will be randomized into two groups using a computer-generated block-of-four randomization sequence. The randomization sequence was generated by independent support staff and concealed using sequentially numbered opaque envelopes. The investigator allocated patients by opening the corresponding envelope to determine group assignment, either to receive the Thoracolumbar interfascial plane block (TLIP group) or the local anesthetic infiltration (LA group). Anesthesiologists, nurses in the Post Anesthesia Care Unit (PACU) and the orthopedic ward staff were blinded to the group allocations.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- LA Group (Active Comparator): Local anesthetic infiltration (0.25%marcaine 40 ml)
  Interventions: Procedure: Local anesthetic infiltration
- TLIP Group (Experimental): Thoracolumbar interfascial plane block with 0.25%marcaine 40 ml under USG
  Interventions: Procedure: Thoracolumbar interfascial plane block

INTERVENTIONS:
Procedure: Thoracolumbar interfascial plane block — Ultrasound-guild bilateral Thoracolumbar interfascial plane block with a total 40 ml, 0.25% bupivacaine by anesthesiologist
  Arms: TLIP Group
Procedure: Local anesthetic infiltration — 0.25%bupivacaine infiltration at surgical wound site by orthopedic surgeon
  Arms: LA Group

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of the thoracolumbar interfascial plane block (TLIP block) versus local anesthetic (LA) infiltration in managing postoperative pain in minimally invasive surgery (MIS) for spine surgery.

The primary outcome was total morphine consumption. Secondary outcomes included pain scores using the the numerical verbal scale (NRS), opioid-related side effects, time of the first request for rescue analgesia, time to ambulation and hospital length of stay.

DETAILED DESCRIPTION:
A single-center, prospective, double-blind, randomized controlled trial at Queen Savang Vadhana Memorial Hospital.

All 40 enrolled patients were randomized to receive the assigned intervention, Thoracolumbar interfascial plane group (TLIP group) and local anesthetic (LA) infiltration group (LA group).

* For TLIP group, patients will receive ultrasound-guild bilateral TLIP block with a total of 40 ml of 0.25% Bupivacaine.
* For LA group, patients will receive local anesthetic infiltration with a same drug by orthopedic surgeon.

At the end of surgery, patients were extubated and transferred to the PACU before being shifted to the orthopedic ward.

Postoperative assessments began upon admission to the PACU, designated as time zero, and continued at regular intervals in the orthopedic ward (6-, 8-, 12- and 24-hours post-surgery).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* American Society of Anesthesiologists classes I-III
* Able to use a patient-controlled analgesia (PCA) device
* Able to rate their pain using a numerical verbal scale (NRS)

Exclusion Criteria:

* Declined to participate
* Uncooperative or unable to complete study assessments
* Had contraindications to the medications used in the study protocol and regional anesthesia.
* History of alcohol or substance abuse within two years prior to surgery,
* Allergies to medication used in the study protocol
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-25 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours
  Total doses of morphine requirement during first 24 hours postoperative period (The investigators recorded at 6,8,12 and 24 hours, postoperatively)

SECONDARY OUTCOMES:
Pain score (NRS) | 24 hours
  The investigators recorded pain score at 6,8,12, 24 hours postoperatively. The scale ranges from 0 to 10, where 0 represents the lowest score and 10 represents the highest score
Postoperative nausea and vomiting | 24 hours
  The investigators recorded the occurrence of postoperative nausea and vomiting (PONV) as present or absent.
Length of hospital stay | 2 weeks
  The investigators recorded the number of hospital days from admission to discharge.
Time of the first request for rescue analgesia | 24 hours
  Time when a patient first asks for pain relief after their surgery.
Respiratory depression | 24 hours
  The investigators recorded the occurrence of respiratory depression as present or absent.

CONTACTS AND LOCATIONS:
Overall Officials: Sophitnapa Tanasittiboon, Anesthesiologist, Study Director — Queen Savang Vadhana Memorial Hospital, Thailand
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Chon Buri, Changwat Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: No